CLINICAL TRIAL: NCT06784102
Title: Clinical Assessment of Pain Levels and Debonding Forces Using the Damon Clear Debonding Plier: a Split-mouth Controlled Clinical Trial
Brief Title: Clinical Evaluation of Pain and Debonding Forces with Damon Clear Debonding Plier Utilizing a Third Wedging Arm
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Baghdad (Other)
Responsible Party: Principal Investigator, Layth Nissan, Assistant Proffessor, University of Baghdad
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: 606422
Record Dates: First submitted 2025-01-10; First posted 2025-01-20 (Actual); Last update posted 2025-01-20 (Actual); Status verified 2021-01

CONDITIONS: Pain Intensity Assessment
Keywords: debonding pain; debonding forces; Damon clear debonding plier; Bracket remover plier; Force-sensitive plier prototype

STUDY DESIGN:
Intervention Model Description: This study employs a split-mouth approach, where each patient undergoes two different interventions: one side of the mouth is treated using the traditional bracket remover plier (control), while the other side is treated using the Damon clear debonding plier (intervention). This design minimizes variability by allowing direct comparison of outcomes (pain levels and debonding forces) within the same individual.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Bracket debonding plier group (No Intervention): The control group (n=40 subjects) involved brackets debonding on the right side (upper and lower quadrants from central incisor to second premolar) of each patient, utilizing a bracket remover debonding plier
- Damon clear debonding plier group (Experimental): The study group B (n=40) encompassed debonding on the left side (upper and lower quadrants from central incisor to second premolar) of each patient, employing the Damon clear debonding plier
  Interventions: Other: Damon Clear Debonding Plier (the primary intervention being tested in this study).

INTERVENTIONS:
Other: Damon Clear Debonding Plier (the primary intervention being tested in this study). — This clinical trial evaluates two types of orthodontic debonding pliers: the Damon Clear Debonding Plier and the traditional Bracket Remover Debonding Plier. The Damon Clear plier features a third wedging arm, which applies an additional lingual or palatal force in addition to the standard occluso-gingival force. The study is designed to assess and compare pain levels and debonding forces between the two pliers. A total of 40 patients, aged 17-25, were treated with both devices using a split-mouth design. The Damon Clear Plier is tested on one side of the mouth while the Bracket Remover Plier is used on the opposite side. Pain perception was measured immediately after the debonding procedure using the Numerical Rating Scale (NRS), and the forces applied during debonding were measured with a force-sensitive prototype. The study aims to identify the device that provides effective debonding with less pain.
  Arms: Damon clear debonding plier group

SUMMARY:
This clinical study aimed to assess pain levels and debonding forces using two different pliers: the traditional bracket remover plier and the Damon clear debonding plier. A total of 40 orthodontic patients (ages 17-25) participated in a split-mouth controlled trial. The patients were divided into two groups, with Group A (Control) using the traditional bracket remover plier and Group B using the Damon clear plier, which features a third wedging arm. Pain perception was evaluated using the Numerical Rating Scale (NRS), and debonding forces were measured using a force-sensitive prototype.

DETAILED DESCRIPTION:
This clinical assessment of pain levels and debonding forces using the Damon clear debonding plier was designed as a split-mouth controlled trial to evaluate the efficacy and comfort of two orthodontic debonding methods. Pain is a significant concern during orthodontic treatment, often influencing patient compliance and overall satisfaction. While research has focused extensively on pain during active treatment, less attention has been directed toward discomfort associated with the removal of orthodontic brackets. Debonding, an integral step in concluding orthodontic treatment, should ideally be painless and harmless to the enamel. However, the discomfort experienced by patients during this process remains a largely underexplored domain. This study sought to fill this gap by comparing pain levels and debonding forces between two types of pliers: the traditional bracket remover plier and the Damon clear debonding plier, the latter featuring a third wedging arm.

The study included 40 orthodontic patients aged 17 to 25 years who had completed comprehensive treatment with metallic brackets. A split-mouth design was utilized, where the right side of each patient's mouth, including the upper and lower quadrants from the central incisor to the second premolar, was treated using the traditional bracket remover plier, categorized as Group A. The left side of the mouth, comprising the same set of teeth, was treated with the Damon clear debonding plier, categorized as Group B. Each plier was modified with a strain gauge load cell and connected to a digital weighting indicator scale, creating a force-sensitive prototype capable of precisely measuring the forces applied during debonding.

Participants were screened for eligibility based on strict inclusion and exclusion criteria to ensure standardization. Inclusion criteria required patients to have a full set of permanent teeth (excluding third molars), no significant dental restorations, no psychological conditions, and an ability to comprehend and respond to anxiety and pain assessment questionnaires. Patients with missing teeth, craniofacial abnormalities, mobile teeth, or a history of recent medications that could influence pain perception were excluded. Prior to the procedure, participants' anxiety levels were assessed using two validated tools: the Generalized Anxiety Disorder Assessment (GAD-7) and the Modified Dental Anxiety Scale (MDAS). Those with high anxiety scores were omitted to avoid potential bias.

Pain perception was measured immediately after the debonding procedure using the Numerical Rating Scale (NRS), chosen for its reliability and preference among patients. The force applied during bracket removal was recorded for each tooth. The debonding process targeted the first five teeth in each quadrant, ensuring uniformity in the procedure. A blinded statistician analyzed the collected data using the T-test, with statistical significance set at p<0.05.

ELIGIBILITY:
Inclusion Criteria:

* individuals aged 17-25 years with the ability to comprehend and respond to questionnaires
* no recent medication intake
* the presence of all permanent teeth except third molars
* sound teeth with minimal prior dental interventions
* brackets bonded with 3M bonding agent and composite (3M, St. Paul, U.S)
* no debonded brackets at the time of assessment
* completion of orthodontic treatment using upper and lower fixed appliances with metallic brackets (Roth/MBT prescription, Dentaurum, Ispringen, Germany,)
* absence of miniscrews at the completion of treatment

Exclusion Criteria:

* patients who were unable to understand the questionnaires,
* those with missing teeth (excluding third molars)
* teeth with prostheses
* craniofacial deformities affecting dentoalveolar bone
* previous surgeries
* heavily restored teeth
* mobile teeth
* teeth with endodontic fillings
* cases with ceramic or plastic brackets
* patients with psychological problems or under psychological medication

Ages: 17 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes — males and females
Enrollment: 40 (Actual)
Dates: Start 2022-01-15 (Actual); Primary Completion 2023-07-15 (Actual); Study Completion 2023-07-15 (Actual)

PRIMARY OUTCOMES:
pain level estimation | Time frame was immediate, as pain perception was assessed immediately after debonding. Pain levels were measured using a Numerical Rating Scale (NRS) right after the procedure to capture the immediate discomfort and pain
  discomfort or pain experienced by patients during the removal of orthodontic brackets from their teeth, patients were prompted to assign a numerical rating scale (NRS) score, ranging from 0 to 10, to assess the perception of pain associated with each individual bracket and the corresponding tooth

SECONDARY OUTCOMES:
debonding forces | Time frame was immediate, as the force required to detach the brackets was measured immediately during the debonding procedure using a force-sensitive plier prototype, which recorded the force at the exact moment of bracket detachment
  the amount of force required to detach an orthodontic bracket from a tooth during the debonding process. It is an important factor in determining the effectiveness and safety of the procedure. Excessive debonding force can cause damage to the enamel or surrounding tissues, while insufficient force may lead to a delay or incomplete removal of the brackets. The force is typically applied through specific tools (debonding pliers), and the direction and distribution of the force can influence both the ease of brackets removal and the potential for patient discomfort

CONTACTS AND LOCATIONS:
Locations (1):
- University of Baghdad, College of Dentistry, Baghdad, Iraq

IPD SHARING:
Plan to Share IPD: No
confidentiality of research and participants information

REFERENCES:
- See also: Patients' report of discomfort and pain during debonding of orthodontic brackets: a comparative study of two methods — https://pubmed.ncbi.nlm.nih.gov/21490985/